CLINICAL TRIAL: NCT04704037
Title: Mobilizing Early Management of Mental Health Complications After Mild Traumatic Brain Injury
Acronym: M4
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Noah Silverberg, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H20-00562
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Concussion
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Minimally enhanced usual care (Active Comparator): See intervention/treatment description
  Interventions: Other: Generic information about concussion management
- Arm 2: Guideline implementation tool (Experimental): See intervention/treatment description
  Interventions: Other: Guideline implementation tool

INTERVENTIONS:
Other: Guideline implementation tool — Family physicians will receive a tailored letter with their patient's mental health screening test results and associated mental health treatment recommendations from the Ontario Neurotrauma Foundation guidelines, as well as a list of mental health treatment resources. In addition, the patient will receive a written information package about mental health problems after mTBI and treatment options to discuss with their family physician.
  Arms: Arm 2: Guideline implementation tool
Other: Generic information about concussion management — Family physicians will receive a generic letter drawing their attention to Canadian clinical practice guidelines for mild Traumatic Brain Injury (developed by the Ontario Neurotrauma Foundation). Patients will receive instructions about how to access generic education materials about mTBI (from concussion.vch.ca/), which they should have received anyway as part of usual care.
  Arms: Arm 1: Minimally enhanced usual care

SUMMARY:
Mental health problems frequently complicate recovery from mild traumatic brain injury (mTBI) but are under-recognized and under-treated. Our research program aims to identify evidence-based strategies for closing this knowledge-practice gap. Building on a successful pilot trial, the reseachers will evaluate the effectiveness of a clinical practice guideline implementation tool designed to support proactive management of mental health complications after mTBI in primary care.

DETAILED DESCRIPTION:
Goal: To determine if a clinical practice guideline implementation tool, designed to support proactive management of mental health complications, can improve clinical outcomes from mild traumatic brain injury (mTBI).

Background: Up to 1 in 4 people who sustain an mTBI develop depression or an anxiety disorder within the first 3 months. Mental health problems triple the risk of long-term disability after mTBI. However, mental health disorders after mTBI are under-detected and under-treated. Canadian clinical practice guidelines for mTBI developed by the Ontario Neurotrauma Foundation (ONF) recommend that family physicians proactively screen and initiate treatment for mental health disorders.

Aims: To evaluate the effectiveness of an implementation intervention designed to facilitate timely detection and treatment of mental health complications in primary care.

Approach: Triple-blinded (treatment provider, patient, assessor) cluster randomized controlled trial with two arms. The intervention involves collecting screening test results from patients and a complex intervention with two components: sharing the screening test results in an actionable format with their family physician and activating patients for the clinical encounter with the family physician by sharing education materials about mental health problems and treatment options after mTBI. The comparison group is usual care.

Hypotheses: The researchers hypothesize that the guideline implementation tool will be associated with lower rates of mental health complications at 26 weeks post-injury, compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-69 years old,
* presentation to emergency department within 72 hours of injury,
* probable mTBI diagnosis per emergency department chart review and interview based on World Health Organization Neurotrauma Task Force diagnostic criteria,
* fluent in English,
* primary residence in British Columbia,
* designate a specific family physician or walk-in clinic where they plan to seek follow-up care

Exclusion Criteria:

* Pre-existing unstable/serious medical condition (e.g., cancer, multiple sclerosis, etc.)
* Pre-existing unstable/severe mental illness (e.g., schizophrenia requiring hospital admission in past year)

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 537 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
MINI version 7.0.2 for DSM-5 | 26 weeks post injury
  Structured diagnostic interview

SECONDARY OUTCOMES:
Rivermead Postconcussion Symptom Questionnaire | 2, 12, 26 weeks post injury
  Standardized questionnaire
World Health Organization Disability Assessment Schedule 2.0 12-item version | 12 and 26 week post injury
  Standardized interview

CONTACTS AND LOCATIONS:
Overall Officials: Noah Silverberg, Principal Investigator — University of British Columbia
Locations (9):
- Canada (9):
  - Urgent and Primary Care Center: North Vancouver, North Vancouver, British Columbia
  - Lion's Gate Hosital, North Vancouver, British Columbia
  - University Hospital of Northern British Columbia, Prince George, British Columbia
  - Richmond Hospital, Richmond, British Columbia
  - Mount Saint Joseph's Hospital, Vancouver, British Columbia
  - Vancouver General Hospital, Vancouver, British Columbia
  - University of British Columbia Hospital, Vancouver, British Columbia
  - Urgent and Primary Care Center: City Center, Vancouver, British Columbia
  - St. Paul's Hospital, Vancouver, British Columbia

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request
Supporting Information: Study Protocol, ICF
Time Frame: October 2025

REFERENCES:
- [Derived] Mikolic A, Snell DL, Theadom A, Faulkner JW, Zemek R, Silverberg ND. The prognostic value of a screening tool for psychological risk factors after mild traumatic brain injury: prospective studies in Canada and New Zealand. BMJ Open. 2025 Sep 10;15(9):e089471. doi: 10.1136/bmjopen-2024-089471. PMID 40935420
- [Derived] Kashyap I, Silverberg ND, Mikolic A. Gender Differences in Seeking and Receiving Healthcare After Mild Traumatic Brain Injury. J Head Trauma Rehabil. 2025 Nov-Dec 01;40(6):469-478. doi: 10.1097/HTR.0000000000001085. Epub 2025 Nov 4. PMID 40705783
- [Derived] Silverberg ND, Rioux M, Mikolic A, Perez DL, Burke MJ, Howard A. Somatic Symptom Disorder After Mild Traumatic Brain Injury. J Head Trauma Rehabil. 2026 Jan-Feb 01;41(1):E18-E26. doi: 10.1097/HTR.0000000000001068. Epub 2025 Dec 29. PMID 40384095
- [Derived] Silverberg ND, Otamendi T, Brasher PM, Brubacher JR, Li LC, Lizotte PP, Panenka WJ, Scheuermeyer FX, Archambault P; Canadian Traumatic Brain Injury Research Consortium (CTRC). Effectiveness of a guideline implementation tool for supporting management of mental health complications after mild traumatic brain injury in primary care: protocol for a randomised controlled trial. BMJ Open. 2022 Jun 21;12(6):e062527. doi: 10.1136/bmjopen-2022-062527. PMID 35728892